CLINICAL TRIAL: NCT02288767
Title: The Effect of Fluid Management by SVV of FloTrac/ Vigileo™ Monitoring on Postoperative Recovery in Bowel Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2014-0730
Record Dates: First submitted 2014-11-03; First posted 2014-11-11 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Bowel Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): For the traditional method group, crystalloid and colloid (maximum 50 ml/kg) are provided through the traditional method of assessing the blood pressure, heart rate and urine volume.
  Interventions: Device: Conventional arterial blood pressure monitoring
- SVV group (Experimental): The method of fluid administration to be employed (traditional or SVV via a FloTrac/ EV1000™ monitor) is determined based on the group. Fluid administration is performed in accordance with the group; in general, about 10 ml/kg/h is administered although it may vary for each patient depending on the preoperative fasting, fluid loss during surgery (evaporation, emanation, urination, surgical area, etc.), and blood loss. Crystalloid is administered in the SVV-monitored group with a target below SVV 12%, and a 200-300 ml of colloid (maximum 50 ml/kg) is loaded when SVV is above 12%. If the patient shows hypertension even when SVV is below 12%, a vasoconstrictor should be administered intermittently or consistently.
  Interventions: Device: Stroke volume variation monitoring with arterial blood pressure monitoring

INTERVENTIONS:
Device: Conventional arterial blood pressure monitoring
  Arms: Control group
Device: Stroke volume variation monitoring with arterial blood pressure monitoring
  Arms: SVV group

SUMMARY:
During an enterectomy, especially in an open surgery, large amounts of fluid are administered in consideration of the patient's fasted state, maintaining blood pressure during surgery and potential third space loss. However, it has recently been reported that excessive fluid administration during surgery is actually detrimental to patients' prognoses. In fact, several reports have suggested that compared to limited fluid administration, excessive fluid administration increased the length of stay or the chances of complications. Thus, goal-directed fluid optimization is required during surgery because only a proper amount of fluid (neither limited nor excessive) administration can minimize postoperative complications and enhance prognosis. In general, the amount of fluid administered is determined with regard to the patient's volume status, including a comprehensive assessment of vital signs such as the pulse rate and blood pressure, and urine volume. However, this method has limitations in that it is an inadequate indicator of the actual intravascular volume of a patient to determine and administer the proper amount of fluid. Recently, new methods of measuring volume status that are less invasive and more accurate have been introduced. These methods include stroke volume variation (SVV) that monitors changes in arterial pressure waveform amplitudes with regard to breathing patterns. This is an effective method of monitoring fluid responsiveness after placing a catheter via a radial artery puncture. The stroke output is dependent on the preload, afterload, and cardiac contractility. The cardiac output is determined by multiplying the stroke output and heart rate. SVV indicates the difference in stroke output within one breathing cycle. A direct or indirect measurement of stroke output is required, which can be performed by analyzing arterial pressure waveforms via a FloTrac Sensor (Edwards Lifesciences, USA) monitor. SVV is known to have a high fluid responsiveness even during open surgeries, yet there is practically no research data on its effect in patients' postoperative recovery and prognosis in comparison to the traditional methods of fluid administration. Therefore, the investigators will apply SVV via a FloTrac/ Vigileo™ monitor on patients undergoing bowel resection to determine whether it better assists proper fluid administration compared to the traditional method of fluid administration by examining the patients' postoperative prognosis such as bowel movement recovery and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 70 scheduled to undergo bowel resection open surgery below the ASA class 3

Exclusion Criteria:

* Patients with significant impairments in heart, kidney, and liver functions
* Patients with arrhythmia such as tachycardia and atrial fibrillation or patients on pacemakers
* Patients diagnosed with peripheral arterial disease or are Allen's test positive
* Patients who underwent surgery on the identical surgical area
* Patients with obesity
* Patients with blood coagulation impairments

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Recovery of bowel movement - gas passing time after bowel resection | 24 hous
  To evaluate the difference in bowel movement recovery whether using SVV or not on the fluid management in the patients undergoing open enterectomy, the difference of postoperative gas passing time will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, College of Medicine, Yonsei Health System, Yonsei Cancer Center, Seoul, South Korea